CLINICAL TRIAL: NCT05775211
Title: Effects of Intrauterine Administration of Autologous Peripheral Blood Mononuclear Cells (PBMC) Modulated With Interferon Tau (IFNt) on Endometrial Cell Populations
Brief Title: Effects of Intrauterine Administration of Autologous PBMC Modulated With IFNt on Endometrial Cell Populations
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nadezhda Women's Health Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7/28022023
Record Dates: First submitted 2023-03-07; First posted 2023-03-20 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Infertility
Keywords: intrauterine PBMC; interferon tau; endometrium; endometrial cell populations; window of implantation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: All participants will undergo the same procedures.
Masking Description: Data analysis will be performed by investigators blind to the biopsy group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Endometrial composition before and after autologous modulated PBMC administration (Experimental): The endometrial cell composition in terms of cell quantities and spatial distribution will be compared before and after intrauterine administration of immunomodulated PBMC.
  Interventions: Biological: Intrauterine administration of PBMC immunomodulated with IFNt

INTERVENTIONS:
Biological: Intrauterine administration of PBMC immunomodulated with IFNt — Standard density gradient centrifugation will be performed to obtain autologous PBMC from patients' peripheral blood (9 ml). Isolated cells will be suspended in RPMI 1640 supplemented with 10% HSA (human serum albumin) and incubated in the presence of 500 IU/ml IFNt for 24 h at 37˚C. The cultured cell suspension will be introduced into the uterine cavity via a catheter.

SUMMARY:
The aim of this clinical trial is to investigate the change in endometrial composition during the window of implantation following intrauterine administration of PBMC immunomodulated with IFNt.

Patients seeking assisted reproductive therapy will be invited to participate. Two endometrial biopsies will be obtained from each patient during mid-secretory phase of two consecutive menstrual cycles. The first biopsy will be obtained one month before the intervention, and the second one - a day after intrauterine administration of the tested cell treatment which will take place the following month.

Immunohistochemistry analysis of the cell composition of the endometrium will be performed.

DETAILED DESCRIPTION:
Female patients with no known uterine pathologies and good general health undergoing treatment for unexplained infertility will be identified and invited to participate in the study. Endometrial biopsy will be obtained seven days after luteinizing hormone (LH) surge during a natural cycle. The following month, 5 days after LH surge, peripheral blood mononuclear cells (PBMC) will be isolated from patients' peripheral blood by density gradient (1.077g/ml) centrifugation and suspended in culture medium. The obtained PBMC will be incubated with 500 IU IFNt at 37˚C for 24 hours. This cell suspension will be carefully introduced in the uterine cavity by catheter on day 6 post LH surge. A second biopsy will be obtained the following day (LH+7).

Immunohistochemistry evaluation of endometrial tissue will be performed in terms of quantities and spatial distribution of various cell types.

ELIGIBILITY:
Inclusion Criteria:

* Participating in Assisted Reproduction Treatment
* Having primary infertility
* Having regular menstrual cycles
* Having signed informed consent

Exclusion Criteria:

* Uterine pathologies
* Endometrial bacterial infections
* Active endometrial inflammation
* Polycystic ovary syndrome
* Presence of auto antibodies such as anti-TPO (thyroid peroxidase), anti-TG (thyroglobulin), ACA (anticentromere antibodies), APA (antiphospholipid antibodies), ANA (antinuclear antibodies), and anti-dsDNA
* Presence of mutations involving the coagulation system such as deficiency of factor XII, Pro C, Pro S
* Oncological condition
* Positive HIV (human immunodeficiency virus), HCV (hepatitis C virus) or HBV (hepatitis B virus) tests

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-03-14 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Change in the numbers of certain endometrial cell populations (immune cells, stem cells, senescent cells) from their levels one month prior to intrauterine administration of immunomodulated PBMC | One month prior to and one day following intrauterine administration of cell treatment
  Immunohistochemical analysis of endometrial biopsies

CONTACTS AND LOCATIONS:
Locations (1):
- Nadezhda Women's Health Hospital, Sofia, Sofia, Bulgaria

IPD SHARING:
Plan to Share IPD: No